CLINICAL TRIAL: NCT06241040
Title: Effects of Aerobic Exercise With and Without Core Muscle Strengthening on Pain, Menstrual Pattern and Quality of Life in Endometriosis
Brief Title: Effects of Aerobic Exercise and Core Muscle Strengthening on Pain, Menstrual Pattern and QOL in Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S22C14G92019
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Endometriosis
Keywords: Endometriosis; Menstrual pattern; Aerobic Exercise; Core Muscle Strengthening; Quality of Life
MeSH Terms: conditions — Endometriosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group with Core Muscle strengthening Group (Experimental): Participants assigned to this group will undergo a combination of aerobic exercise and core muscle strengthening interventions. The aerobic exercise component will be similar to the first group, while additional exercises targeting the core muscles (abdomen, back, and pelvis) will be included.
  Interventions: Other: Aerobic Exercises with core Muscle strengthening
- Aerobic Exercise without Core Muscle Strengthening Group (Active Comparator): Participants assigned to this group will engage in aerobic exercise interventions
  Interventions: Other: Aerobic Exercise without Core Muscle Strengthening

INTERVENTIONS:
Other: Aerobic Exercises with core Muscle strengthening — Participants assigned to this group will undergo a combination of aerobic exercise and core muscle strengthening interventions. The aerobic exercise component will be similar to the first group, while additional exercises targeting the core muscles (abdomen, back, and pelvis) will be included.
  Arms: Aerobic Exercise Group with Core Muscle strengthening Group
Other: Aerobic Exercise without Core Muscle Strengthening — Aerobic Exercise without Core Muscle Strengthening
  Arms: Aerobic Exercise without Core Muscle Strengthening Group

SUMMARY:
Endometriosis is a complex and debilitating gynecological condition affecting millions of women worldwide. It is characterized by the abnormal growth of endometrial-like tissue outside the uterus, leading to chronic pelvic pain, dysmenorrhea, dyspareunia, and reduced quality of life. While pharmacological interventions are commonly prescribed to manage symptoms, their efficacy may be limited, and they often come with adverse effects. Therefore, exploring non-pharmacological approaches, such as exercise, is crucial in improving the management of endometriosis-related symptoms. Aerobic exercise has gained attention as a potential therapeutic intervention for endometriosis due to its positive effects on pain modulation, hormonal regulation, and overall well-being.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will be conducted at Jinnah Hospital in Lahore, Pakistan, to investigate the effects of aerobic exercise with and without core muscle strengthening on pain, menstrual pattern, and quality of life in women diagnosed with endometriosis. The study will employ a convenient randomization sampling technique, aiming to recruit approximately 30 participants who meet the inclusion criteria. Eligible participants will be reproductive-age women experiencing endometriosis-related pain, with regular menstrual cycles or irregularities associated with endometriosis. They should be medically stable, cleared for physical activity, and willing to participate in an exercise intervention program. Exclusion criteria include pregnancy, severe endometriosis-related complications, significant comorbidities, recent surgery, ongoing hormonal treatments targeting endometriosis, inability to participate in exercise programs, and severe mental health conditions. By investigating these interventions, the study seeks to improve symptom management, menstrual regularity, and overall quality of life for women with endometriosis while considering safety and feasibility within the study setting.

Keywords: Endometriosis, Menstrual pattern, Aerobic Exercise, Core Muscle Strengthening, Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with endometriosis.(16)
* Age range (e.g., 18-49 years)
* Regular menstrual cycles or menstrual irregularities associated with endometriosis.
* Medically stable and cleared for participation in physical activity.
* No contraindications for aerobic exercise or core muscle strengthening

Exclusion Criteria:

* Pregnant individuals or those actively trying to conceive.
* Recent endometriosis-related surgeries/procedures
* Use of hormonal therapies/medications targeting endometriosis
* Severe endometriosis complications requiring immediate medical intervention
* Inability to engage in aerobic exercise.
* Significant cardiovascular/respiratory conditions
* Concurrent participation in another exercise/rehabilitation program

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Endometriosis occur during Menstrual Cycle
Enrollment: 30 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Pain: | 8 weeks
  The Visual Analog Scale (VAS) for Pain is a commonly used instrument for assessing pain intensity. It is a subjective measure that asks individuals to rate their pain on a continuous line or scale. The VAS typically consists of a 10 cm line with anchor points representing "no pain" on one end and "worst possible pain" on the other end. Participants are instructed to mark the line at the point that represents their current level of pain.
Endometrial Health Profile-30 Endometrial Health Profile | 8 weeks
  The EHP-30 (Endometrial Health Profile-30) is a specific questionnaire designed to assess the impact of endometriosis on various aspects of a person's life. It is a self-report instrument that measures health-related quality of life in individuals with endometriosis.
Menstrual pattern Bleeding score MIQ questionnaire | 8 weeks
  The Menstrual Pattern Bleeding Score MIQ (Menstrual Impact Questionnaire) questionnaire is a specific tool used to assess the impact of menstrual patterns and bleeding on individuals' lives. It is a self-report questionnaire that measures the severity and impact of menstrual symptoms and irregularities on various aspects of daily functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Taufiq, PPDPT, Principal Investigator — Riphah International University, Senior Lecturer
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No